CLINICAL TRIAL: NCT02976922
Title: Characterisation of the Salivary and Faecal Microbiome in Patients With Recurrent Aphthous Stomatitis Before and After Treatment With Probiotics
Brief Title: The Salivary and Faecal Microbiome of Recurrent Aphthous Stomatitis Patients Before and After Treatment With Probiotics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Anne Marie Lynge Pedersen, Associate Professor, PhD, DDS, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-15012527
Record Dates: First submitted 2016-02-07; First posted 2016-11-30 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Recurrent Aphthous Ulcers
Keywords: RAS; microbiome; probiotics
MeSH Terms: conditions — Stomatitis, Aphthous

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic lozenge (Active Comparator): Probiotic lozenge, one lozenge twice daily for 3 months. The lozenge contains Lactobacilli Reuteri (100 billions colony forming units (CFU)/tablet)
  Interventions: Dietary Supplement: Probiotic lozenge
- Placebo (Placebo Comparator): Placebo lozenge, one lozenge twice daily for 3 months
  Interventions: Dietary Supplement: Probiotic lozenge

INTERVENTIONS:
Dietary Supplement: Probiotic lozenge — 10 patients with RAS are randomised to active treatment with probiotic lozenge, one lozenge twice daily for 3 months and other 10 patients with RAS are randomised to treatment with placebo lozenge, one lozenge twice daily for 3 months.
  Other Names: Biogaia

SUMMARY:
Recurrent aphthous stomatitis (RAS) is one of the most common ulcerative diseases affecting the oral mucosa. The aetiology remains unknown, but several local, systemic, immunologic, genetic, allergic, nutritional, and microbial factors have been proposed as causative agents. Clinically, RAS is characterised by recurrent bouts of one or several rounded, shallow, painful oral ulcers at intervals of a few months or days. The aim of this study is to characterise the salivary and faecal microbiome in 20 patients with RAS and compare the findings with those of 20 healthy controls. The study also includes a double-blind randomized placebo-controlled intervention with probiotics (Lactobacillus reuteri-containing lozenges 2 tablets daily for 3 months) or placebo. The salivary and faecal microbiome in RAS patients is compared before and after treatment. This study will improve our understanding of the pathogenesis in RAS and provide us with knowledge on potential future therapeutic approaches.

DETAILED DESCRIPTION:
Purpose of the study The purpose of this study is to characterise the salivary and faecal microbiome in patients with recurrent aphthous stomatitis (RAS) and to compare the findings to those of a matched healthy control group. Another purpose is to investigate the effect of treatment with probiotics on the microbiome in whole saliva and faeces as well as the severity and number of RAS outbreaks. Moreover, a smear will be taken from present aphthous ulcers before and after treatment with probiotics in order to characterise the local microbiota.

It is assumed that the microbiome in whole saliva and faeces from patients with RAS (minor or major type aphthous ulcers) differs from the microbiome in whole saliva and faeces from age- and gender-matched control persons.

It is also hypothesised that probiotic treatment has a beneficial effect on the mucosal pain and reduces the severity of RAS and the frequency of outbreaks. Furthermore, it is assumed that treatment with probiotic has an effect on microbiome in whole saliva and faeces from patients with RAS.

Background Recurrent aphthous stomatitis (RAS) is one of the most common ulcerative diseases affecting the oral mucosa. The prevalence varies from 5-25%. The aetiology remains unknown, but several local, systemic, immunologic, genetic, allergic, nutritional, and microbial factors have been proposed as causative agents.

Clinically, RAS is characterised by recurrent bouts of one or several rounded, shallow, painful oral ulcers at intervals of a few months or days.

RAS can be classified into three different types: minor, major and herpetiform. Minor RAS comprises about 80% of the cases. This type is characterised by aphthous ulcers with a diameter of about 5 mm, often localised in the buccal and labial mucosa. The ulcers heal within 7-10 days without formation of scars. Major RAS appear in 10-15% of the patients. The ulcers are often crateriform with a diameter of 10-30 mm, and typically present on the labial mucosa, the soft palate, the tonsillar region and oropharynx. The healing time may vary from 2 to 6 weeks and leaving cicatrix. These ulcers are very painful and food intake may be compromised. The prevalence of the herpetiform type is 5-10%.

This type is often localised in the floor of the mouth and the ventral part of the tongue, and it characterised by aggregation of multiple small ulcers.

The aetiology remains unknown, but a number of local and systemic factors are assumed increase the predisposition, including mucosal trauma, stressful events, hormonal changes, smoking cessation, allergy to various food substances as well as vitamin- and/or mineral deficiency. The is also a genetic predisposition as the possibility of developing RAS is 90% if both parents have RAS and 20% if one of the parents has RAS.

Microbial factors A number of microorganisms have been suggested involved in the aetiopathogenesis of RAS. These include oral streptococci, especially Streptococcus mitis, but the cross-reaction between oral streptococci and oral mucosal antigens is unspecific and considered clinically insignificant. Helicobacter pylori, which is associated with gastritis and duodenal ulcers may also be seen in dental plaque and therefore also be suggested involved in the pathogenesis of RAS, but the anti-H. pylori seropositivity has not been found increased in patients with RAS. Various vira have been found in biopsies from aphthous ulcers such as cytomegalovirus and Epstein-Barr virus. Herpes simplex, varicella zoster and adenovirus have also been assumed to play a role in the aetiopathogenesis. However, it is has not been possible to show a causal relationship between virus infection and RAS, and viral DNA may be present due to a secondary infection.

Novel technologies improve our ability to make more in depth analyses of the microbiota in patients with RAS. While working on this study protocol one study on the microbiome in patients with RAS has been published showing an increased proportion of Bacteroides species in the oral mucosa of patients with RAS compared to healthy controls. Thus, as previous studies also suggest the oral microbiota appears to play a role in the development of RAS as well as in perpetuation of RAS.

In this study we will characterise the microbiome in whole saliva, faeces and the aphthous ulcers of patients with RAS (with active lesions) and analyse how it differs from the microbiome of healthy subjects. This characterisation could be essential for our understanding the pathogenesis of RAS and contribute to the development of novel strategies for managing these patients.

Immunopathological factors Several studies indicate that the pathogenesis of RAS includes a number of cell-mediated mechanisms, but the exact immunopathogenesis is still not clarified. Phagocytic and cytotoxic T-lymphocytes may be a role in the destruction of the oral epithelium and the presence of these immune cells is regulated and maintained by local release of cytokines. Patients with outbreak of RAS have an increased presence of gamma-delta T-cells in the blood compared to healthy control persons and patients without active RAS. Moreover, patients with RAS have an increased presence of Tumour Necrosis Factor (TNF)-alpha compared to those who do not have RAS, but also other proinflammatory cytokines like interleukin-2 and -6 are likely to play a role in the pathogenesis of RAS. Finally, aphthous-like ulcers have been found associated to a number of inflammatory bowel diseases such as ulcerative colitis and Crohn's disease and celiac disease as well as cyclic neutropenia, HIV-infection and immunoglobulin A (IgA)-deficiency. Accordingly, an immune component may be involved in RAS which contribute to a change in the intestinal microbiota or vice versa. In this study, we will characterise the microbiota in saliva and in faeces from patients with RAS before, during and after treatment with probiotics.

The study design and methods The project comprises a cross-sectional study which investigates the microbiome in whole saliva and faeces from 20 patients with RAS and 20 healthy control persons. The project also includes a double-blind randomized placebo-controlled intervention with probiotics (Lactobacillus reuteri-containing lozenges 2 tablets daily for 3 months) or placebo. The salivary and faecal microbiome in RAS patients is compared before and after treatment.

The patients with RAS are recruited among patients referred to the Oral Medicine Clinic, Faculty of Health and Medical Sciences, University of Copenhagen. The 20 healthy controls are recruited via www.forsoegsperson.dk

Methods include:

* Interview re. onset of RAS, oral symptoms (assessed by means of a visual analogue scale), comorbidity, medication intake, smoking and alcohol habits, oral hygiene habits.
* Collection of chewing paraffin-stimulated whole saliva.
* Oral examination including evaluation of aphthous ulcers (Ulcer Severity Score), registration of dental status and periodontal status.
* A smear from one of the aphthous ulcers.
* A faecal sample will be collected by the subjects themselves in their homes after thorough instruction and handled according to manual from the Statens Serum Institut. From the sample 250 mg is collected and kept in a freezer kept at -80°C until further processing and analysis.
* A blood test including haemoglobin (HgB), C reactive protein (CRP), iron, cobalamin, folate, transferrin, ferritin and vitamin D levels.

Extraction of bacterial DNA from saliva, faecal and smear samples (at baseline, 7-day and 90-day of intervention with probiotics or placebo, respectively) will be carried out in the laboratory at Department of Odontology, University of Copenhagen, using previously established procedures based on instructions from the Human Microbiome Project.

Metagenomic analyses on extracted bacterial DNA from saliva, smear and faecal samples are made by Beijing Genomics Institute. Illumina 16S rDNA sequencing allows determination of bacterial taxonomy and phylogenetic diversity.

ELIGIBILITY:
Inclusion criteria

* Patients with recurrent aphthous stomatitis (minor or major aphthous ulcers) and Caucasians
* Healthy and non-medicated subjects who match the patients with regard to age and gender

Exclusion Criteria:

* Autoimmune diseases/immunosuppressive conditions
* Treatment with immunosuppressant
* Current treatment with antibiotics
* Drug and/or alcohol abuse
* Pregnancy
* Current use of oral rinses
* Current use of topical steroids or other agents for relief oral symptoms

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Beneficial effect of probiotics on the size of aphthous ulcers and the frequency of RAS outbreaks | 3 months
  Measurements of the size and numbers of aphthous ulcers (in mm, using scoring system) Baseline (Day 0), Day and after 30 days
Beneficial effect of probiotics on oral pain related to aphthous ulcers | 3 months
  Visual analogue pain scale (0-100 mm) Baseline (Day 0), Day 7 and after 30 days

SECONDARY OUTCOMES:
Changes in salivary and faecal microbiome in patients with RAS due to use of probiotics | 3 months
  Baseline (Day 0), Day 7 and after 30 days: Bacterial DNA extraction and metagenomic analyses on saliva, ulcer smear and faeces

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine Bukkehave, Scholarstip, Principal Investigator — Department of Odontology, University of Copenhagen; Eric Bennett, Assoc Prof, Principal Investigator — Department of Odontology, University of Copenhagen
Locations (1):
- Department of Odontology, University of Copenhagen, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pedersen AML, Bukkehave KH, Bennett EP, Twetman S. Effect of Lozenges Containing Lactobacillus reuteri on the Severity of Recurrent Aphthous Ulcers: a Pilot Study. Probiotics Antimicrob Proteins. 2020 Sep;12(3):819-823. doi: 10.1007/s12602-019-09586-x. PMID 31410765